CLINICAL TRIAL: NCT02430259
Title: Effectiveness and Tolerability of Weekly Rifapentine/Isoniazid for 3 Months for Tuberculosis Preventive Treatment: A Randomized Controlled Study in China
Brief Title: Efficacy of Weekly Rifapentine and Isoniazid for Tuberculosis Prevention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 81373064
Record Dates: First submitted 2015-04-16; First posted 2015-04-30 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Silicosis; Tuberculosis
Keywords: rifapentine; isoniazid; QuantiFERON Gold In-Tube; tuberculin skin test
MeSH Terms: conditions — Silicosis; Tuberculosis | interventions — Isoniazid; rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weekly Isoniazid / Rifapentine (Experimental): Weekly INH / RRT given by DOT
  Interventions: Drug: Weekly INH / RRT given by DOT
- No preventive treatment (No Intervention): Follow up without intervention

INTERVENTIONS:
Drug: Weekly INH / RRT given by DOT — weekly oral Rifapentine 15 mg/kg (up to 900mg) plus Isoniazid 15 mg/kg (up to 900mg) for 12 doses
  Other Names: isoniazid; I; INH; rifapentine; RPT; 3 RPT/INH
  Arms: Weekly Isoniazid / Rifapentine

SUMMARY:
Tuberculosis (TB) remains the most important infectious disease in the world. Preventive treatment plays an important role in successful control of TB. For preventive therapy, the three-month (12-dose) regimen of weekly rifapentine and isoniazid (3RPT/INH) are now recommended by WHO for its non-inferiority, safety and convenience compared with 6~9 months regimen of daily isoniazid monotherapy or 3~4 months daily rifampicin monotherapy. And the treatment completion rate is higher compared with daily regimen. However, relevant study is lacking in China where the TB burden is high with the incidence rate of 70/100, 000. And the provision of chemoprophylaxis is not recommended in China currently.

Silicosis is a high risk factor of Mycobacterium tuberculosis infection. This is an open-label, randomized, Phase III clinical trial to evaluate the effectiveness and tolerability of the 3RPT/INH to prevent tuberculosis (TB) compared with those who do not receive preventive treatment among silicotic patients.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains the most important infectious disease in the world. Preventive treatment plays an important role in successful control of TB. For preventive therapy, the three-month (12-dose) regimen of weekly rifapentine and isoniazid (3RPT/INH) are now recommended by WHO for its non-inferiority, safety and convenience compared with 6~9 months regimen of daily isoniazid monotherapy or 3~4 months daily rifampicin monotherapy. And the treatment completion rate is higher compared with daily regimen. However, relevant study is lacking in China where the TB burden is high with the incidence rate of 70/100, 000.

Silicosis is a high risk factor of Mycobacterium tuberculosis infection. This is an open-label, randomized, Phase III clinical trial to evaluate the effectiveness and tolerability of the 3RPT/INH to prevent tuberculosis (TB) among silicotic patients.

The PRIMARY objective of this open-label, randomized, Phase III clinical trial is to evaluate the effectiveness of the 3RPT/INH to prevent TB compared with those who do not receive preventive treatment among eligible silicotic patients.

The SECONDARY objective:

Describe the safety profile of 3RPT/INH in China (the rates of drug discontinuation for any reason and due to adverse drug reactions associated with 3RPT/INH, the rates of any grade 3, 4, or 5 drug toxicity associated with 3RPT/INH) Describe the treatment completion rates of 3RPT/INH. Describe patterns of antibiotic resistance of M. tuberculosis isolates in patients who develop TB despite preventive treatment.

Compare the results of QuantiFERON Gold In-Tube before and after preventive treatment.

For assessment of the primary outcome, development of TB, a sample size of approximately 280 persons per arm will be required with 3 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Silica exposure or diagnosed with silicosis;
* Age between 18 to 65 years;
* Willing to provide signed informed consent, or parental consent and participant assent.

Exclusion Criteria:

* Clinical or culture confirmed active TB;
* A history of treatment for > 14 consecutive days with a rifamycin or > 30 consecutive days with INH during the previous 2 years;
* A documented history of a completing an adequate course of treatment for active TB or latent TB infection;
* Allergy to Isoniazid, Rifampin, or Rifapentine;
* Human immunodeficiency virus (HIV) infection;
* History of hepatitis B/C infection or liver cirrhosis;
* Serum Aspartic transaminase (AST) or alanine transaminase (ALT) > 2x upper limit of normal or total bilirubin >2.5 mg/dL;
* Receiving immunosuppressants or biological agents;
* Life expectancy <3 years;
* Mental disorder;
* Participated in other clinical trials in recent three months;
* Other conditions that investigates consider not suitable for participate.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Cumulative rate of culture-confirmed or clinically diagnosed TB disease in participants | 3 years

SECONDARY OUTCOMES:
Percentage of participants with drug discontinuation for any reason and due to adverse drug reactions associated with 3RPT/INH | up to 30 days after the last dose of study drug
Percentage of patients with Grade 3 or 4 drug toxicities and deaths associated with 3RPT/INH | up to 30 days after the last dose of study drug
Percentage of participants who complete the treatment regimen | Enrollment up to Month 3 (3RPT/INH)
The proportion of rifampicin and/or isoniazid resistance of M. tuberculosis isolates in patients who develop TB in preventive treatment group. | 3 years
Measure the quantitative and qualitative changes of the results of QuantiFERON Gold In-Tube before and after preventive treatment. | Enrollment up to 3 months after preventive treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, MD,PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Wenling No.1 People's Hospital, Zhejiang, Taizhou, Zhejiang, China

REFERENCES:
- [Derived] Xu H, Zhou J, Yang Q, Yang Y, Zhou F, Qian M, Lin X, Zhang W, Shao L, Ruan Q. QuantiFERON-TB supernatant-based biomarkers predicting active tuberculosis progression. Int J Infect Dis. 2025 Aug;157:107915. doi: 10.1016/j.ijid.2025.107915. Epub 2025 May 3. PMID 40320069
- [Derived] Ruan QL, Yang QL, Gao YX, Wu J, Lin SR, Zhou JY, Shao LY, Wang S, Liu QQ, Gao Y, Jiang N, Zhang WH. Transcriptional signatures of human peripheral blood mononuclear cells can identify the risk of tuberculosis progression from latent infection among individuals with silicosis. Emerg Microbes Infect. 2021 Dec;10(1):1536-1544. doi: 10.1080/22221751.2021.1915184. PMID 34042560
- [Derived] Ruan QL, Huang XT, Yang QL, Liu XF, Wu J, Pan KC, Shen YJ, Cai LM, Ling Q, Jiang T, Hong JJ, Wang XD, Ma CL, Peng GQ, Wang XZ, Mao JC, Wu TZ, Lin MY, Shao LY, Zhang WH. Efficacy and safety of weekly rifapentine and isoniazid for tuberculosis prevention in Chinese silicosis patients: a randomized controlled trial. Clin Microbiol Infect. 2021 Apr;27(4):576-582. doi: 10.1016/j.cmi.2020.06.008. Epub 2020 Jun 15. PMID 32553881
- [Derived] Yang Q, Ruan Q, Liu X, Shen Y, Jiang T, Wu J, Cai L, Pan K, Lin M, Huang X, Shao L, Zhang W. Preventive tuberculosis treatment effect on QuantiFERON TB-Gold in-tube testing in a high tuberculosis-endemic country: A clinical trial. Int J Infect Dis. 2020 Feb;91:182-187. doi: 10.1016/j.ijid.2019.11.023. Epub 2019 Nov 23. PMID 31770617